CLINICAL TRIAL: NCT03876652
Title: Effect of Pacemaker With Closed Loop Sensor on Quality of Life and Recurrence of Syncope in Patients With Neuromodulated Syncope Refractory to Medical Treatment: Randomized Double-blind Clinical Trial
Brief Title: Pacemaker Effect With Closed Loop Sensor in Neuromodulated Syncope Refractory to Medical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Mauricio Duque Ramirez, Mauricio Duque, CES University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 719
Record Dates: First submitted 2019-01-14; First posted 2019-03-15 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Syncope
Keywords: Syncope; Presyncope; Time; Vasovagal; Unconsciousness
MeSH Terms: conditions — Syncope; Unconsciousness

STUDY DESIGN:
Intervention Model Description: Prospective, multi-institutional, randomized, double-blind intervention study. Patients with a diagnosis of cardioinhibitory syncope will be included. They have implanted a pacemaker with a closed loop sensor. Pacemakers are left in CLS mode during the first month, the month in the implant is cited patients and the random form is left reprogrammed in DDD-R or DDD-CLS mode as randomization is established. After 4 months of this last visit, the reprogramming mode will be exchanged and left for another 4 months. During this time, a clinical and electrophysiological evaluation will be performed. At the end of these 8 months, the patient will be rescheduled in the same electrophysiologist's mode as the patient has felt better. The clinical follow-up will continue for 12 more months. At the end of the study, the results of the quality of life scales will be analyzed, the occurrence of episodes of syncope, the reduction of pre-syncopal symptoms, mode and programming will be evaluated.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DDD-CLS (Experimental): Patients with a pacemaker programmed in DDD-CLS mode
  Interventions: Device: Pacemaker with Closed Loop Stimulation (CLS)
- DDD-R (Active Comparator): Patients with a pacemaker programmed in DDD-R mode
  Interventions: Device: Pacemaker with Closed Loop Stimulation (CLS)

INTERVENTIONS:
Device: Pacemaker with Closed Loop Stimulation (CLS) — In active mode of closed loop sensor (CLS), evaluate its impact on quality of life and recurrence of syncope.

SUMMARY:
Vasovagal syncope is an entity frequently in the emergency services, its treatment includes pharmacological and non-pharmacological measures, and in some severe cases, requires the implantation of cardiac stimulation devices, specifically, those pacemakers that have closed-loop sensors (CLS).

This research is an intervention study, multi-institutional, randomized and double blind that will be carried out in patients older than 18 years, with a diagnosis of neurally mediated type 1, 2A or 2B syncope documented in a tilting table test, who have had at least 2 syncope in the last year and that significantly affects the quality of life despite the use of pharmacological and non-pharmacological non-interventionist therapy.

This study aims to evaluate the effect of cardiac pacing therapy with CLS pacemakers on quality of life, recurrence of syncope and pre-syncopal symptoms in patients with a diagnosis of neurally mediated syncope in this group of patients.

DETAILED DESCRIPTION:
Syncope is defined as a loss of consciousness with inability to maintain the postural tone, with subsequent spontaneous recovery and without neurological sequelae. This occurs due to cerebral hypoperfusion by two mechanisms: 1) decreased cardiac output, usually due to bradycardia, and 2) hypotension due to decreased peripheral vascular resistance. An incidence of 6.2 per 1000 persons / year has been calculated, constitutes 2% of the reasons for consultation by emergency department and is found in 40% of the hospitalized participants. Its prevalence increases with age and is clearly influenced by the presence or absence of heart disease. The most frequent etiology is vasovagal, which has a benign course, with a mortality that does not exceed the expected for the general population. However, up to 21.6% have recurrences, which affects the quality of life and can generate physical injuries, especially in the geriatric population. The pathophysiology is not completely clear, it is thought that orthostasis has an important mechanism by decreasing the venous return, therefore, this leads to a vigorous contraction of the myocardium in the presence of a little filled heart chamber, it can stimulate the mechanoreceptors and thus precipitate the Bezold Jarisch reflex, which results in paradoxical hypotension and bradycardia.

The management can be variable, and will depend on the patient's response, from conservative strategies such as changes in lifestyle, avoiding triggers, abortive maneuvers in the case of prodromes, and some drugs (fludrocortisone) to cardiac stimulation devices such as pacemakers. Cardiac stimulation has been studied in participants with cardioinhibitory response in the Tilt test with divergent results, especially with the use of conventional pacemakers that monitor the fall in heart rate. Interestingly, an other type of pacemakers, those with closed handle sensor (CLS), that measures the impedance through each beat, which is related to myocardial contractility, in this way it could detect changes in the contractility that precede the cardioinhibitory response, and thus guarantee a good cardiac output and avoid syncope.

The use of cardiac stimulation therapy has been proposed as an effective strategy in participants with recurrent syncope and refractory to pharmacological and non-pharmacological measures, a special group are those with a cardioinhibitory response with asystole greater than 6 seconds, however, this benefit it could be extrapolated to those of mixed commitment. In the world, there is no definitive consensus on the level of recommendation for the implantation of pacemakers with CLS in this disease, however, based on the pathophysiology, studies of the disease and technical elements on the functioning of these devices, they have come implanting in Colombia and in the world with apparent good results in the quality of life of the participants, syncope-free event rate, longer time to the first syncope and improvement in hemodynamic parameters in the Tilt Test. In Colombia, more research is needed to confirm or reject this assertion.

General objective: Evaluate the effect of cardiac pacing therapy with CLS pacemakers on quality of life, recurrence of syncope and pre-syncopal symptoms of participants with a diagnosis of neurally mediated syncope (with mixed response or inhibitory cardio) refractory to pharmacological and non-pharmacological management, in six health care centers in the city of Medellín.

Specific objectives

* Sociodemographically and clinically characterize the study population.
* Evaluate the impact on quality of life, pre and post implant.
* Measure the occurrence of episodes of syncope, pre and post implant.
* Assess the reduction of pre-syncopal symptoms.
* Evaluate if the mode and programming functions influence the appearance of syncopes and recurrences.
* Determine the average time that elapses from the implantation of the CLS pacemaker until the first episode of syncope.

Interventions of participants

* A: participants who will be activated the CLS function one month after implantation of the pacemaker. They will be reevaluated after 4 months and will be changed to DDD-R mode for another 4 months, when the results will be analyzed to define the final form of reprogramming.
* B: patient to whom, one month after the implantation of the pacemaker, the R function will be activated. They will be reevaluated after 4 months and will be switched to DDD-CLS mode for another 4 months, when they will be evaluated again and the results will be analyzed for define final form of reprogramming.

Participants will be contacted through the electrophysiology service of "CES Cardiology" in Medellín, Colombia.

The calculation of the sample size was carried out probabilistically with the following parameters and based on the previous studies: Power 80%, confidence: 95%, expected proportion of group 1: 72%, expected proportion group2: 99% What gave the following results: intervention A: 26 participants, intervention B: 26 participants. Total sample: 52 participants.

Selection of participants All participants will be recruited and who meet all the inclusion criteria and none of the exclusion criteria will be selected by one of the members of the research team previously trained on the Plan of Clinical Research and that has been designated to perform this type of tasks.

Estimated time to include participants The inclusion of all participants requires approximately 6 months. The anticipated duration of this study is 27 months. This will depend on the inclusion rate.

Informed consent process: It will be prepared by the principal investigator, with the information indicated in article 15 of resolution 8430.

* It will be reviewed by the Human Research Ethics Committee of the CES University and can only be signed by the patient, researchers and witnesses when it is approved.
* Indicate the names and contact forms of the principal investigators and who should be contacted in case of any difficulty or adverse event.
* It must be signed by two witnesses and by the research subject or his legal representative. If the research subject does not know how to sign, he will print his fingerprint and in his name he will sign another person that he designates.
* It will be prepared in duplicate, leaving a copy in the possession of the research subject or his legal representative.

Blinding of the study: The programming modes of the intracardiac devices can only be known through the use of specific reprogramming equipment provided by each generating company of the device. In the case of pacemakers with CLS, their only manufacturer is Biotronik, so they provide a device that connects with the device that the patient has implanted. Unless the reprogramming card is delivered, neither the patient nor another person will be able to establish the programming mode.

In this way the people who will be in contact with the programming of the device will be:

Electrophysiologist in charge of implanting the device: it could be any of the members of the CES Cardiology group with this training, it will implant the device and leave it in DDD-CLS mode to start the first month or washing time. This electrophysiologist will not make any scheduled visits or reprogram the device in any of his visits.

Electrophysiologist commissioned the visit by electrophysiology within each of the visits scheduled and listed above: professional in charge of programming the devices as established by the paper envelopes generated in the random assignment. It will be the only person who will know the way of programming during the 8 months of intervention and will not disclose this information to the patient or their relatives.

Main co-investigators: they will not know the way of programming the device nor will they attend the part of the visit that performs electrophysiology. In another office and before or after the program, they will evaluate the patient clinically and ask the questions included in the scales of quality of life used.

The person who will analyze the information: will know the process. The patient: He will not know the programming mode of his device, that is, he will not know if he is in DDD - CLS or DDD - R. This study will be double blind.

Random assignment Through computer-based randomization programs, 26 participants will be assigned to the group of participants who, in the month of implantation, will be programmed in DDD-CLS mode and 26 participants who will be programmed in DDD-R mode one month after implantation. The randomization will be known by the investigating epidemiologist who will activate the randomization program and the electrophysiologist who will program the patient. Initial randomized programming modes will be delivered in sealed envelopes to the electrophysiologist who will program the patient.

Procedures The clinical trial will be conducted in accordance with the Clinical Research Plan. All those who participate in the conduct of the clinical study will be qualified by training, training or experience to carry out their tasks and this training should be documented in an appropriate manner. The clinical study will not begin until it receives written approval from the Ethics Committee and the relevant regulatory authorities and all necessary documentation has been collected. Procedures during the time of intervention. Once the patient enters the health center with criteria to participate in the study, as long as it does not meet any of the exclusion criteria and has signed the informed consent (the participant or a legal representative in case this is not in conditions to sign).

Starting point: Prior to implanting the device. Between the day of implantation and the first month (at which time the initial visit will take place) will be the washing or "wash out" process in which the device will be left in DDD-CLS mode until the start visit.

Start visit: One month after implanting the device. It includes two parts: Evaluation by electrophysiology and Clinical evaluation.

Visit # 1: It will happen 4 months after the start visit. It includes two parts: Evaluation by electrophysiology and Clinical evaluation.

Visit # 2: Finally, a final check (visit # 2) will be made 8 months after the start visit and 4 months after the visit # 1. It includes two parts: Evaluation by electrophysiology and Clinical evaluation.

Procedures during the time following the end of the intervention: At the end of the 8 months in which the information on the mode of reprogramming was recorded and these modes were reversed, the follow-up will continue for 12 more months counted from visit # 2 as follows:

* Visit # 3: It will take place 6 months after the visit # 2 and 14 months after the initial visit. The patient will be evaluated clinically (without pacemaker programming) by one of the researchers who will apply the SFSQ and SF-36 quality of life scales.
* Visit # 4: It will take place 12 months after the visit # 2 and 20 months after the initial visit. The patient will be evaluated clinically (without pacemaker programming) by one of the researchers who will apply the SFSQ and SF-36 quality of life scales.

After this the study ends.

Procedures in case of Adverse Events: In the event of any adverse event related or not to the implant or use of the device or any condition of the patient, the patient must notify the group of researchers in the contact telephone numbers that are delivered and according to the severity and needs of the event will be cited in an additional visit for clinical evaluation and / or electrophysiology or will be redirected to the CES Clinic if the event or situation requires management in the emergency department or intrahospital service. Each of these adverse events must be reported on a form and a communication sent within 72 hours after the group of researchers had knowledge of the Human Research Ethics Committee of the CES University, making the event known to all. the details.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Diagnosis of neurally mediated syncope with a tilting table test (Tilt test) that demonstrates a mixed (type 1) or cardioinhibitory response (Type 2A and 2B).
* Negative impact on work and social life.
* Non-respondent to pharmacological therapy (Fludrocortisone 0.1mg / 24 hours for 3 months) and non-pharmacological (exercise, hydration and consumption of more than 3 months) is due to a cardiologist who has performed a strict stricture over time.
* At least 2 episodes of syncope in the last year.

Exclusion Criteria:

* Complete atrioventricular block.
* Second degree ventricular atrial block.
* Bradycardia syndrome - tachycardia.
* Disease of the sinus node.
* Arrhythmia (bradycardia or tachycardia that generate syncope and / or low cardiac output).
* Syncope due to hypersensitivity of the carotid sinus.
* Syncope with Tilt Test that demonstrates depressant vasopressor response (type 3).
* Refusal of the patient, his relatives or the attending physician to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in the quality of life with pacemaker CLS with Syncope Functional Status health-related quality of life Questionnarie (SFSQ). | 21 months
  To evaluate the results of pacemaker therapy with pacemaker with CLS in the quality of life, the score of the scales is compared: SFSQ of implanting the pacemaker, a statistical analysis with tests is performed paired.
  The quality of life questionnaire consists of several domains consisting of questions that evaluate the parameters of daily life with multiple-choice questions with a single answer. At the end of the questionnaire, each question in its domain of a score and once each domain has a representation in the final qualification.
Change in the quality of life with pacemaker CLS with the score Short Form - 36 (SF-36). | 21 months
  To evaluate the results of pacemaker therapy with pacemaker with CLS in the quality of life, the score of the scales is compared: SF-36 (Short form - 36) of implanting the pacemaker, a statistical analysis with tests is performed paired.
  The quality of life questionnaire consists of several domains consisting of questions that evaluate the parameters of daily life with multiple-choice questions with a single answer. At the end of the questionnaire, each question in its domain of a score and once each domain has a representation in the final qualification.
Change of number of syncopes | 21 months
  Change in the number of syncopes with the use of CLS pacemakers in participants with neuromediated syncope

SECONDARY OUTCOMES:
Change in free time of syncope | 21 months
  The use of CLS pacemaker increases the time until the first episode of syncope occurs in participants with neurally mediated syncope
Presence or absence of pre-syncopal symptoms: postural dizziness | 21 months
  The use of CLS pacemaker improves postural dizziness in participants with neurally mediated syncope ( (will ask at the clinic visit before completing the quality of life questionnaires).
Presence or absence of pre-syncopal symptoms: fatigue | 21 months
  The use of CLS pacemaker improves fatigue in participants with neurally mediated syncope (will ask at the clinic visit before completing the quality of life questionnaires).
Presence or absence of pre-syncopal symptoms: headache | 21 months
  The use of CLS pacemaker improves headache in participants with neurally mediated syncope (will ask at the clinic visit before completing the quality of life questionnaires).
Presence or absence of pre-syncopal symptoms: sleep disturbance | 21 months
  The use of CLS pacemaker improves sleep disturbance in participants with neurally mediated syncope (will ask at the clinic visit before completing the quality of life questionnaires).
Presence or absence of pre-syncopal symptoms: alterations in temperature. | 21 months
  The use of CLS pacemaker improves alterations in temperature in participants with neurally mediated syncope (will ask at the clinic visit before completing the quality of life questionnaires).

OTHER OUTCOMES:
Demographic characteristics | 21 months
  Describe the demographic characteristics of the participants.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - CES Cardiología sede Sandiego, Medellín, Antioquia
  - Clínica CES, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet analyzed the possibility of sharing or not sharing these data.

REFERENCES:
- [Background] Linzer M, Pontinen M, Gold DT, Divine GW, Felder A, Brooks WB. Impairment of physical and psychosocial function in recurrent syncope. J Clin Epidemiol. 1991;44(10):1037-43. doi: 10.1016/0895-4356(91)90005-t. PMID 1940996
- [Background] van Dijk N, Sprangers MA, Boer KR, Colman N, Wieling W, Linzer M. Quality of life within one year following presentation after transient loss of consciousness. Am J Cardiol. 2007 Aug 15;100(4):672-6. doi: 10.1016/j.amjcard.2007.03.085. Epub 2007 Jun 26. PMID 17697827
- [Background] Goyal P, Maurer MS. Syncope in older adults. J Geriatr Cardiol. 2016 Jul;13(5):380-6. doi: 10.11909/j.issn.1671-5411.2016.05.002. No abstract available. PMID 27594863
- [Background] Blanc JJ. Syncope: Definition, Epidemiology, and Classification. Cardiol Clin. 2015 Aug;33(3):341-5. doi: 10.1016/j.ccl.2015.04.001. PMID 26115819
- [Background] Rosanio S, Schwarz ER, Ware DL, Vitarelli A. Syncope in adults: systematic review and proposal of a diagnostic and therapeutic algorithm. Int J Cardiol. 2013 Jan 20;162(3):149-57. doi: 10.1016/j.ijcard.2011.11.021. Epub 2011 Dec 20. PMID 22188993
- [Background] Bassetti CL. Transient loss of consciousness and syncope. Handb Clin Neurol. 2014;119:169-91. doi: 10.1016/B978-0-7020-4086-3.00013-8. PMID 24365296
- [Background] van Dijk N, Sprangers MA, Colman N, Boer KR, Wieling W, Linzer M. Clinical factors associated with quality of life in patients with transient loss of consciousness. J Cardiovasc Electrophysiol. 2006 Sep;17(9):998-1003. doi: 10.1111/j.1540-8167.2006.00533.x. Epub 2006 Jun 9. PMID 16764705
- [Background] Occhetta E, Bortnik M, Audoglio R, Vassanelli C; INVASY Study Investigators. Closed loop stimulation in prevention of vasovagal syncope. Inotropy Controlled Pacing in Vasovagal Syncope (INVASY): a multicentre randomized, single blind, controlled study. Europace. 2004 Nov;6(6):538-47. doi: 10.1016/j.eupc.2004.08.009. PMID 15519257
- [Background] Russo V, Rago A, Papa AA, Golino P, Calabro R, Russo MG, Nigro G. The effect of dual-chamber closed-loop stimulation on syncope recurrence in healthy patients with tilt-induced vasovagal cardioinhibitory syncope: a prospective, randomised, single-blind, crossover study. Heart. 2013 Nov;99(21):1609-13. doi: 10.1136/heartjnl-2013-303878. Epub 2013 May 30. PMID 23723446
- [Background] Connolly SJ, Sheldon R, Roberts RS, Gent M. The North American Vasovagal Pacemaker Study (VPS). A randomized trial of permanent cardiac pacing for the prevention of vasovagal syncope. J Am Coll Cardiol. 1999 Jan;33(1):16-20. doi: 10.1016/s0735-1097(98)00549-x. PMID 9935002
- [Background] Sutton R, Ungar A, Sgobino P, Russo V, Massa R, Melissano D, Beiras X, Bottoni N, Ebert HH, Francese M, Jorfida M, Giuli S, Moya A, Andresen D, Brignole M; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Cardiac pacing in patients with neurally mediated syncope and documented asystole: effectiveness analysis from the Third International Study on Syncope of Uncertain Etiology (ISSUE-3) Registry. Europace. 2014 Apr;16(4):595-9. doi: 10.1093/europace/eut323. Epub 2014 Jan 9. PMID 24406537
- [Background] Brignole M. International study on syncope of uncertain aetiology 3 (ISSUE 3): pacemaker therapy for patients with asystolic neurally-mediated syncope: rationale and study design. Europace. 2007 Jan;9(1):25-30. doi: 10.1093/europace/eul135. PMID 17224418
- [Background] Brignole M, Menozzi C, Moya A, Andresen D, Blanc JJ, Krahn AD, Wieling W, Beiras X, Deharo JC, Russo V, Tomaino M, Sutton R; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Pacemaker therapy in patients with neurally mediated syncope and documented asystole: Third International Study on Syncope of Uncertain Etiology (ISSUE-3): a randomized trial. Circulation. 2012 May 29;125(21):2566-71. doi: 10.1161/CIRCULATIONAHA.111.082313. Epub 2012 May 7. PMID 22565936
- [Background] Palmisano P, Zaccaria M, Luzzi G, Nacci F, Anaclerio M, Favale S. Closed-loop cardiac pacing vs. conventional dual-chamber pacing with specialized sensing and pacing algorithms for syncope prevention in patients with refractory vasovagal syncope: results of a long-term follow-up. Europace. 2012 Jul;14(7):1038-43. doi: 10.1093/europace/eur419. Epub 2012 Jan 13. PMID 22247273
- [Background] Lindovska M, Kamenik L, Pollock B, Hoenen S, Bokelmann T, Spitzer W, Salbach P, Behroz A, Frey A. Clinical observations with Closed Loop Stimulation pacemakers in a large patient cohort: the CYLOS routine documentation registry (RECORD). Europace. 2012 Nov;14(11):1587-95. doi: 10.1093/europace/eus062. Epub 2012 Mar 28. PMID 22455935
- [Background] Occhetta E, Bortnik M, Vassanelli C; INVASY Italian Feasibility Study Group. The DDDR closed loop stimulation for the prevention of vasovagal syncope: results from the INVASY prospective feasibility registry. Europace. 2003 Apr;5(2):153-62. doi: 10.1053/eupc.2002.0292. PMID 12633640
- [Background] Bortnik M, Occhetta E, Dell'Era G, Secco GG, Degiovanni A, Plebani L, Marino P. Long-term follow-up of DDDR closed-loop cardiac pacing for the prevention of recurrent vasovagal syncope. J Cardiovasc Med (Hagerstown). 2012 Apr;13(4):242-5. doi: 10.2459/JCM.0b013e328351daf5. PMID 22367575
- [Background] Kanjwal K, Karabin B, Kanjwal Y, Grubb BP. Preliminary observations on the use of closed-loop cardiac pacing in patients with refractory neurocardiogenic syncope. J Interv Card Electrophysiol. 2010 Jan;27(1):69-73. doi: 10.1007/s10840-009-9452-1. Epub 2009 Nov 25. PMID 19937372
- [Background] Puppala VK, Dickinson O, Benditt DG. Syncope: classification and risk stratification. J Cardiol. 2014 Mar;63(3):171-7. doi: 10.1016/j.jjcc.2013.03.019. Epub 2014 Jan 7. PMID 24405895
- See also: Use of closed loop sensor pacing system in patients with vasovagal syncope refractory to medical treatment — https://doi.org/10.1016/j.rccar.2015.07.012
- See also: Closed Loop Stimulation for Neuromediated Syncope (SPAIN Study) (SPAIN) — https://clinicaltrials.gov/ct2/show/NCT01621464